CLINICAL TRIAL: NCT03834129
Title: Interest of Intravenous Dexmedetomidine (Dexdor®) in the Knee Replacement Surgery Performed Under Locoregional Anesthesia: a Randomized, Double Blind, Controlled Clinical Trial
Brief Title: Dexmedetomidine Intra Venous Arthroplasty
Acronym: DIVA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018/08
Record Dates: First submitted 2019-02-05; First posted 2019-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Primary Total Knee Arthroplasty
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Dex group) intravenous infusion of dexmedetomidine (Experimental): Pre-anesthetic and per-operative intravenous infusions of dexmedetomidine 1µg/kg in 250ml of sodium chloride 0.9%
  Interventions: Drug: Dexmedetomidine
- (Control group) intravenous infusion of physiological serum (Placebo Comparator): Pre-anesthetic and per-operative intravenous infusions of 250ml of sodium chloride 0.9%
  Interventions: Drug: sodium chloride 0.9%

INTERVENTIONS:
Drug: Dexmedetomidine — Two administrations, before anesthesia and during surgery, by intravenous infusion of dexmedetomidine 1 μg/kg in 250 ml of physiological serum for 30 minutes
  Arms: (Dex group) intravenous infusion of dexmedetomidine
Drug: sodium chloride 0.9% — Two administrations, before anesthesia and during surgery, by intravenous infusion of 250 ml of physiological serum for 30 minutes
  Arms: (Control group) intravenous infusion of physiological serum

SUMMARY:
Intravenous dexmedetomidine is a drug used in reanimation with sedative, anxiolytic and sympatholytic properties. Recent studies showed useful properties for anaesthesia : decrease of morphine consumption after a various type of surgery, sedative effect on patients under regional anaesthesia, prolongation of central or peripheral regional block. Dose-ranging study for intravenous dexmedetomidine showed that 2 µg/kg is an effective dose to prolong interscalene block. This study aims to determine if intravenous dexmedetomidine at 2 µg/kg allows a longer analgesic duration after a quadri-block (femoral, subgluteal sciatic, obturator and alateral cutaneous nerve blocks) with ropivacaine 0.32% for total knee replacement under regional anaesthesia.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind controlled trial with two parallel groups. All patients undergoing total knee arthroplasty under regional anaesthesia and sedation will be screened for inclusion in the protocol. In the pre-anaesthesia room, after the implementation of classical monitoring with an oxygen mask and a peripheral venous catheter, all patients will receive an antibioprophylaxy according to SFAR recommendations and injection of 10 mg of IV dexamethasone.

The patients will be then randomized in 2 groups:

* Dexmedetomidine group (Dex group) : Two administrations of 1 microg/kg of Dexdor® in 250 ml of sodium chloride during 30 min. The first injection will be performed in the pre-anaesthesia unit and the second in the operating room with a free interval of 60 min between the beginning of the 2 injections.
* Control group : Two administrations of 250 ml of sodium chloride during 30 min according to the same former recommendations.

Under ultrasonography guidance and with in-plan technic, a quadri-block (femoral, sciatic subgluteal, obturator and lateral cutaneous nerve blocks) with a maximum of 225 mg of ropivacaine diluted in 70 ml of sodium chloride (ropivacaine 0.32 %) will be performed. If needed, sedation with 5 µg of sufentanil and 1 to 2 mg of midazolam will be performed before regional anaesthesia.

In the operating room, under close monitoring, the patients will receive a bolus of Ketamine 0.3 mg/kg and a propofol bolus of 0.3 mg/kg followed by a continuous infusion if needed. The total dose of propofol used for sedation, conversion to general anaesthesia or any complications concerning anaesthesia or dexmedetomidine (hypotension, bradycardia, arrhythmia, advance cardiac block) will be collected. Postoperative analgesia will be reached with IV 1 g paracetamol and 100 mg ketoprofen starting during surgery and following in the surgical ward by oral paracetamol 1 g / 6 h and oral ibuprofen 400 mg / 8 h. In post anaesthesia care unit all the patients will have oxycodone titration if pain VRS (verbal rating scale) >3 and oxycodone 10 mg/ 4 h in the surgical ward if pain VRS (verbal rating scale) >3.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Patients undergoing elective total knee arthroplasty
* Consent for participation
* Affiliation to the french social security system
* For women of child bearing potential without contraception, beta-HCG negative result

Exclusion Criteria:

* Chronic pain syndrome requiring preoperative morphine use (class 3)
* Hypersensitivity to dexmedetomidine
* Allergy to nonsteroidal anti-inflammatory drugs
* Contraindication for locoregional anesthesia
* Patient wishing a general anesthesia
* Weight>100 kg, obstructive sleep apnea syndrome or gastrooesophageal reflux complicating the sedation with spontaneous ventilation
* Known acute ischemic disease
* Severe liver failure
* Uncontrolled low blood pressure
* Heart rate < 60 bpm
* Advanced cardiac block (Level 2 or 3) except if pacemaker
* Pregnant or breastfeeding women
* Communication difficulties or neuropsychiatric disorder
* Patients under protection of the adults (guardianship, curators or safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-01-11 (Actual); Study Completion 2020-01-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of dexmedetomidine infusion 2 μg/kg in pre-anesthesia and operative room, on duration of postoperative analgesia after a knee arthroplasty performed under locoregional anesthesia. | 48 hours
  Duration of analgesia defined as the time between the performance of regional anesthesia and the first dose of rescue analgesia with opioides.

SECONDARY OUTCOMES:
Incidence of hypotension or bradycardia Events. | 48 hours
  Number of complications due to dexmedetomidine (hypotension or bradycardia episodes)
Maximal postoperative pain. | 48 hours
  Pain VRS verbal rating scale ranging from 0 to 10 (0=no pain, 10=worst possible pain)
Postoperative opioids morphine consumption. | 48 hours
  Postoperative cumulated dose of oxynorm (mg)
Dose of hypnotic drug during surgery. | 4 hours
  Total amount of propofol (mg) administered during surgery
Ability to walk | Days 0, 1 and 2
  Distance < 50 m or > 50 m
Quadricep mobilization | Days 0, 1 and 2
  0 : paralysis ; 1 : paresis ; 2 : normal contraction
Foot elevator muscle mobilization | Days 0, 1 and 2
  0 : paralysis ; 1 : paresis ; 2 : normal contraction

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Médipôle Garonne, Toulouse, Haute-Garonne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chassery C, Marty P, Rontes O, Chaubard M, Vuillaume C, Basset B, Merouani M, Marquis C, De Lussy A, Delbos MC, Casalprim J, Bataille B, Naudin C, Ferre F, Delbos A. Total knee arthroplasty under quadruple nerve block with ropivacaine 0.32%: effect of addition of intravenous dexmedetomidine to intravenous dexamethasone on analgesic duration. Reg Anesth Pain Med. 2021 Feb;46(2):104-110. doi: 10.1136/rapm-2020-101749. Epub 2020 Oct 21. PMID 33087480